CLINICAL TRIAL: NCT00004151
Title: Open Label Phase II Study on XR5000 Administered as a 5 Day Infusion in Advanced Non Small Cell Lung Cancer
Brief Title: Acridine Carboxamide in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16991N; EORTC-16991N
Record Dates: First submitted 1999-12-10; First posted 2004-03-15 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — DACA, acridine

INTERVENTIONS:
Drug: acridine carboxamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of acridine carboxamide in treating patients who have advanced non-small cell lung cancer that cannot be treated with surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of acridine carboxamide on objective response, response rate, and duration of response in patients with unresectable, locally advanced, progressive or metastatic non-small cell lung cancer. II. Determine the toxicities and pharmacokinetics of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive acridine carboxamide IV over 24 hours for 5 days. Treatment repeats every 3 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks until disease progression or commencement of another treatment.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven unresectable, locally advanced, progressive or metastatic non-small cell lung cancer Not amenable to curative surgery or radiotherapy No prior first line chemotherapy for metastatic or advanced disease At least 1 bidimensionally measurable target lesion by CT scan No symptomatic brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) SGOT, SGPT, and alkaline phosphatase no greater than 2 times ULN (5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.7 mg/dL Cardiovascular: No ischemic heart disease within the past 6 months Normal 12 lead ECG Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other prior or concurrent malignancy except cone biopsied carcinoma of the cervix or adequately treated basal or squamous cell skin cancer No unstable systemic disease or active uncontrolled infection No psychological, familial, sociological, or geographical condition that could preclude compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 2 weeks since prior major surgery Other: No other concurrent anticancer agents No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1999-09; Primary Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel R. Hanauske, MD, PhD, MBA, Study Chair — Haemato-Onkologische Praxis und Tagesklinik
Locations (8):
- Kaiser Franz Josef Hospital, Vienna, Austria
- Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - CHU de la Timone, Marseille
- Haemato-Onkologische Praxis und Tagesklinik, Munich, Germany
- Italy (2):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- Hospital Universitario 12 de Octubre, Madrid, Spain